CLINICAL TRIAL: NCT07238270
Title: Research on Physical Fitness and Flatfoot in Children
Status: Active, not recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202400647B0
Record Dates: First submitted 2025-08-29; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Flatfoot
Keywords: physical fitness; flatfoot
MeSH Terms: conditions — Flatfoot | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- preschool students: Children aged about 1-6 years from northern Taiwan.
  Interventions: Other: No intervention (observational study)
- primary school students: Children aged about 7-12 years from northern Taiwan.
  Interventions: Other: No intervention (observational study)
- middle school students: Children aged about 13-15 years from northern Taiwan.
  Interventions: Other: No intervention (observational study)
- high school students: Adolescents aged about 16-18 years from northern Taiwan.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational study with no intervention.

SUMMARY:
This study aims to explore the relationship between children's physical fitness and flatfoot. Specifically, it is designed to determine whether fitness levels are linked to the incidence and severity of flatfoot and to explore other possible factors, including genetics, exercise behavior, and body weight.

DETAILED DESCRIPTION:
This study aims to examine the relationship between children's physical fitness and flatfoot. We will recruit a sample of children across different ages, genders, and fitness levels. Physical fitness will be assessed using standardized tests, including body composition, cardiorespiratory endurance, muscle strength, and flexibility. Foot structure and function will be evaluated through arch index and plantar pressure analysis to determine the presence and severity of flatfoot. Background information, such as age, gender, height, weight, exercise habits, and family history, will also be collected.

ELIGIBILITY:
Inclusion Criteria:

-Children aged 1-18 years

Exclusion Criteria:

* Diagnosed with developmental delays
* Diagnosed with neurological disorders
* Presence of other congenital or acquired conditions causing impairments
* Holders of a disability certificate
* History of asthma
* History of heart disease

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 600 children aged 1-18 years from northern Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire Score | Baseline
  Score from a self-designed questionnaire on lifestyle habits and foot-related symptoms. Scale range: higher scores = better habits, fewer symptoms.
Body Fat Percentage | Baseline
  Body fat percentage measured using InBody analyzer. Unit: Percent (%) (lower values indicate better body composition).
Skeletal Muscle Mass | Baseline
  Skeletal muscle mass measured using InBody analyzer. Unit: Kilograms (higher values indicate greater muscle mass).
Cardiorespiratory Endurance | Baseline
  Performance on standardized shuttle run test. Unit: Seconds (shorter time indicates better endurance).
Handgrip Strength | Baseline
  Grip strength measured using digital dynamometer. Unit: Kilograms (higher values indicate greater strength).
Pinch Strength | Baseline
  Pinch force measured with a pinch gauge. Unit: Kilograms (higher values indicate greater strength).
Flexibility Test | Baseline
  Sit and reach distance measured in centimeters. Unit: Centimeters (higher values indicate greater flexibility).
Balance Ability | Baseline
  Time maintaining one-leg stance without support. Unit: Seconds (longer time indicates better balance).
Arch Index | Baseline
  Foot arch index derived from footprint analysis. Unit: Ratio (0.2-0.3 indicates normal arch).
Achilles Tendon Alignment | Baseline
  Deviation angle of Achilles tendon alignment. Unit: Degrees (smaller angles indicate better alignment).

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD, PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan